CLINICAL TRIAL: NCT04622488
Title: The Effect of Diclofenac Potassium Insitu Gel Versus Calcium Hydroxide as Intra-canal Medications on Post-operative Pain and Anti-bacterial Effect in Lower Non Vital Premolars With Symptomatic Apical Periodontitis
Brief Title: The Effect of Diclofenac Potassium Insitu Gel Vs Calcium Hydroxide as Intra-canal Medications on Post-operative Pain and Anti-bacterial Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Mohamed Aboul Azayem, Prinicipal Investegator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-7-2
Record Dates: First submitted 2020-10-28; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Post Operative Pain
Keywords: Calcium Hydroxide; Diclofenac potassium; Intra-canal Medications
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac Potassium (Active Comparator): In the form of insitu gel can be applied as solution or suspension that undergoes gelation after administration.
  Interventions: Drug: Diclofenac Potassium
- Calcium Hydroxide (Experimental)
  Interventions: Drug: Diclofenac Potassium

INTERVENTIONS:
Drug: Diclofenac Potassium — - In the form of Insitu gel system can be applied as solution or suspension that undergoes gelation after administration. Applied once inside the root canal after chemo-mechanical preparation.
  Other Names: Cataflam

SUMMARY:
The aim of this study is to clinically compare the post-operative pain level and antibacterial effect when using the Diclofenac Potassium Insitu gel versus calcium hydroxide as an intra- canal medication in patients with apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years old.
* Males/Females.
* Lower permanent premolars with: Non-Vital pulps. Sensitive to percussion. Negative response to cold pulp tester (ethyl chloride spray1). Apical periodontitis
* Systemically healthy patients (ASA I or II).

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders. (ASA III or IV).

  * History of intolerance to NSAIDS.
  * Patients with two or more adjacent teeth requiring endodontic treatment.
  * Teeth with :
* Association with swelling or fistulous tract.
* Acute or chronic peri-apical abscess. Mobility Grade II or III.
* Pocket depth more than 5mm.
* Previous root canal therapy.
* Non-restorability
* Patients with a contraindication for the use of DFK or those known to be allergic to any of the study medications.eg. Patient with kidney problems.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post operative pain assessed by VAS | 72 hours
  Post-operative pain following chemo-mechanical endodontic treatment will be measured.
  A pain chart using visual analogue scale (VAS) will be used to record the patients' pain levels. The VAS (0-10 scale) consists of a line anchored by two extremes "No pain" and "the worst pain". Patients will be asked to choose the mark that represented their level of pain from 0 to 10. Pain level will be assigned as follow:
  * 0, "no pain"
  * 1-3, "mild pain"
  * 4-6, "moderate pain"
  * 7-10, "severe pain" Using the VAS chart, the patient will choose and record the most appropriate pain rating according to the pain intensity endured.

SECONDARY OUTCOMES:
Antibacterial effectiveness by measuring the bacterial count. | pre-operatively(S1), after chemo-mechanical preparation(S2), and after 1 week(S3).
  The bacterial count method will be used. Once the samples will arrive to the microbiology department, Cairo University, the tubes containing the thioglycolate 14(transport medium) with the paper points will be placed in micro centrifuge and vortexed for 30 sec. One hundred (100) μl aliquots of the vortexed samples will be placed in a new sterile tube containing 1 ml of thioglycolate to obtain 1/10 concentration to assess the microbial load of common aerobes and anaerobes found in each root canal. The effect of the treatment in each group, the initial colonizers (S1), the mechanical preparation (S2) and after the intra-canal medication (S3) will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, El- Manial, Egypt